CLINICAL TRIAL: NCT03058289
Title: A Phase 1/2 Safety Study of Intratumorally Administered INT230-6 in Adult Subjects With Advanced Refractory Cancers
Brief Title: A Phase 1/2 Safety Study of Intratumorally Dosed INT230-6
Acronym: IT-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intensity Therapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IT-01; KEYNOTE KN-A10 (Other: Merck Sharp & Dohme LLC); CA184-592 (Other: Bristol Myers Squibb Company)
Record Dates: First submitted 2017-02-10; First posted 2017-02-20 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Head and Neck Cancer; Squamous Cell Carcinoma; Lymphoma; Pancreatic Cancer; Liver Cancer; Colon Cancer; Lung Cancer; Bile Duct Cancer; Chordoma of Sacrum; Sarcoma
Keywords: Neoplasm; Malignancy; Intratumoral; Intralesional; anti-PD-1 antibodies; Immuno therapy; Dose escalation; Platinum; Intensity Therapeutics; INT230-6; Cisplatin; Vinblastine; PD-1; Vinca; KEYTRUDA®; Pembrolizumab; CTLA-4; Carcinoma; Yervoy; Ipilimumab; Keynote A10; CA184-592
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Lymphoma; Pancreatic Neoplasms; Liver Neoplasms; Colonic Neoplasms; Lung Neoplasms; Bile Duct Neoplasms; Sarcoma; Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12; Carcinoma | interventions — spartalizumab; pembrolizumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: There were 6 cohorts in the escalation portion of the protocol. Five dosed INT230-6 alone and one was combined with pembrolizumab. Cohorts A and B1 treated superficial tumors at a 1:4 ratio of drug to tumor with a low tumor load once per month. Cohort EA was similar to cohort A with INT230-6 every 2 weeks. Cohort EC escalated the total and maximal dose per any one tumor to a ratio of 1:2 & dosed every two weeks. Cohort EC2 explored a drug load ratio of 1:3 and escalated the dose per tumor further. Cohort DEC combined INT230-6 with a fixed amount of pembrolizumab.
  Completed, non-escalation cohorts include 1) monotherapy INT230-6 cohort (EC3) dosed every two weeks 2) INT230-6 in a combination with pembrolizumab (DEC2) and 3) INT230-6 in combination with ipilimumab (FEC). Other specific regimens or combinations of INT230-6 may be designated by the Study Steering Committee.
Masking Description: There were no masking and all patients received INT230-6 treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Monotherapy With >=40% Total Tumor Burden Dosed (Cohorts A1/B1/EA/EC/EC2/EC3) (Experimental): Dosing: >=40% Total Tumor Burden
  A1:INT230-6 injections into only superficial tumors, low starting dose, low concentration per tumor.
  B1:INT230-6 injections into deep tumors, low starting dose, low drug concentration per tumor
  Dosing schedule for A1 and B1 is every 28 days for 5 sessions
  EA:INT230-6 injections into superficial tumors, medium starting dose, low drug concentration per tumor
  EC:INT230-6 injections into superficial or deep tumors, moderately high starting dose, high drug concentration per tumor
  EC2:INT230-6 injections into superficial or deep tumors, high starting dose, moderate drug concentration per tumor, higher number of tumors to be treated per session than EC.
  EC3:INT230-6 injections at fixed maximal dose into superficial or deep tumors, unlimited number of tumors to be treated per session with retreatment once every 9 weeks for two years.
  Dosing schedule for EA, EC, EC2 and EC3 is every 2 weeks for 5 sessions
  Completed Cohorts
  Interventions: Drug: INT230-6
- Monotherapy With <40% Total Tumor Burden Dosed (Cohorts A1/B1/EA/EC/EC2/EC3) (Experimental): Dosing: <40% Total Tumor Burden
  A1:INT230-6 injections into only superficial tumors, low starting dose, low concentration per tumor.
  B1:INT230-6 injections into deep tumors, low starting dose, low drug concentration per tumor
  Dosing schedule for A1 and B1 is every 28 days for 5 sessions
  EA:INT230-6 injections into superficial tumors, medium starting dose, low drug concentration per tumor
  EC:INT230-6 injections into superficial or deep tumors, moderately high starting dose, high drug concentration per tumor
  EC2:INT230-6 injections into superficial or deep tumors, high starting dose, moderate drug concentration per tumor, higher number of tumors to be treated per session than EC.
  EC3:INT230-6 injections at fixed maximal dose into superficial or deep tumors, unlimited number of tumors to be treated per session with retreatment once every 9 weeks for two years.
  Dosing schedule for EA, EC, EC2 and EC3 is every 2 weeks for 5 sessions
  Completed Cohorts
  Interventions: Drug: INT230-6
- INT230-6 Combined With Pembrolizumab (Cohorts DEC/DEC2) (Experimental): DEC: INT230-6 injections every 2 weeks for 5 sessions with the possibility for INT230-6 retreatment into superficial tumors, with addition of anti-PD-1 antibody KEYTRUDA® (pembrolizumab) dosed concurrently starting at Day 1 every 3 weeks for two years for selected cancer types.
  Completed Cohort
  DEC2:INT230-6 per the dosing of cohort EC3 combined with KEYTRUDA® (pembrolizumab) dosed per DEC concurrently starting at Day 1 for selected cancers.
  Completed Cohort
  Interventions: Drug: INT230-6; Biological: anti-PD-1 antibody
- INT 230-6 Combined With Ipilimumab (Cohort FEC) (Experimental): FEC: INT230-6 per the EC3 regimen combined with Yervoy (ipilimumab) dosed concurrently starting at Day 1 every 3 weeks for four treatments for selected cancer types.
  Completed Cohort anti-CTLA-4 antibody: The anti-CTLA-4 antibody will be added concomitantly with INT230-6 as noted in cohort FEC.
  Interventions: Drug: INT230-6; Biological: anti-CTLA-4 antibody

INTERVENTIONS:
Drug: INT230-6 — INT230-6 is clear sterile solution administered by injection directly into the tumor to be treated.
  The product contains a cell permeation agent with cisplatin and vinblastine sulfate at fixed concentrations.
Biological: anti-PD-1 antibody — The anti-PD-1 antibody will be added concomitantly with INT230-6 as noted in cohort DEC and DEC2
  Other Names: pembrolizumab; KEYTRUDA®; MK-3475
  Arms: INT230-6 Combined With Pembrolizumab (Cohorts DEC/DEC2)
Biological: anti-CTLA-4 antibody — The anti-CTLA-4 antibody will be added concomitantly with INT230-6 as noted in cohort FEC
  Other Names: ipilimumab; Yervoy; BMS-734016
  Arms: INT 230-6 Combined With Ipilimumab (Cohort FEC)

SUMMARY:
This study evaluated the intratumoral administration of escalating doses of a novel, experimental drug, INT230-6. The study was conducted in patients with several types of refractory cancers including those at the surface of the skin (breast, squamous cell, head and neck) and tumors within the body such (pancreatic, colon, liver, lung, etc.). Sponsor also tested INT230-6 in combination with anti-PD-1 and anti-CTLA-4 antibodies.

DETAILED DESCRIPTION:
INT230-6 is comprised of 3 agents in a fixed ratio - a cell permeation enhancer and two, potent anti-cancer payloads (cisplatin and vinblastine sulfate). The penetration enhancer facilitates dispersion of the two drugs throughout injected tumors and enables increased diffusion into cancer cells. Nonclinical safety studies showed no findings following drug injection into healthy tissues.

Historically physicians administer the two active drugs comprising INT230-6 by intravenous (IV) infusion to achieve a systemic blood level at the limit of tolerability. The objective is destroy both visible tumors and unseen circulating cancer cells (micro-metastases). Unfortunately, dosing drugs IV delivers only a small amount with a low concentration at the tumor site. This approach especially for late stage cancers is not highly effective and often quite toxic to the patient.

Attempts at direct intratumoral injection with chemotherapeutic agents have not shown the ability to treat the injected tumor, non-injected tumors or micro-metastases. This lack of efficacy for local administration is due possibly to poor dispersion and a lack of cell uptake of the agents.

Due to the use of the novel cell penetration enhancing agent INT230-6 treatment demonstrated strong efficacy in animals having large tumors. The Sponsor's in vivo, non-clinical data shows that INT230-6 thoroughly saturates and kills injected tumors. In addition, the drug induces an adaptive (T-cell mediated) immune response that attacks not only the injected tumor, but non-injected tumors and unseen micro-metastases. Cured animals become permanently immunized against the type of cancer that INT230-6 eliminates.

Clinical trial IT-01 sought to determine the safety and potential efficacy of dosing INT230-6 directly into several different types of cancers. In addition, animal studies showed a strong synergy of INT230-6 with immune modulation agents. Thus, as part of study IT-01 the Sponsor seeks to understand the safety and efficacy of INT230-6 when administered in combination with immuno-therapeutic agents such as antibodies that target Programmed Cell Death (PD-1 or anti-PD-1) and Cytotoxic T-Lymphocyte Associated Protein 4 (CTLA-4 or anti-CTLA-4) receptors.

This study sought to understand whether tumor regression can be achieved, and patient outcomes improved.

ELIGIBILITY:
Inclusion Criteria:

INT230-6 monotherapy Cohorts EC2 and EC3, combination with KEYTRUDA® cohort DEC2 and combination with Yervoy cohort FEC. Where criteria diverge the DEC2 and FEC specific criteria will be noted.

1. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
2. Men and Women > 18 years of age on the day of signing consent.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status < 2; (for pembrolizumab and ipilimumab combinations please see supplements DEC/DEC2 and FEC for ECOG criteria).
4. Populations: INT230-6 will be injected into deep or superficial tumors for subjects with histologically or cytologically confirmed advanced or metastatic cancers; (for pembrolizumab and ipilimumab combinations please see supplements DEC/DEC2 and FEC for Populations).
5. Includes subjects with loco-regional disease that have relapsed/recurred within 6 months of chemo-radiation and who have no standard of care.
6. Subjects with metastatic disease who have failed one or more approved standard therapies, or have no alternate approved therapy available. Failure of all approved therapies that have a modest or marginal impact on survival is not required as long as the treating physician believes that treatment on study is appropriate for the subject and documents that the subject elects to defer the approved therapies.

   Note: There is no limit on the number of prior therapies that a patient (subject) may have received prior to enrollment in any cohort.
7. Subjects must have measurable disease by iRECIST 1.1 criteria including one target tumor for injection by the local site investigator/radiology. Superficial tumors must have one tumor greater than or equal to 1.0 cm, deep tumors greater than or equal to 1.0 cm (as measured by caliper (for non-injected tumors only) or image guidance). Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Subjects must have a minimum of one injectable lesion as determined by the investigator (for superficial tumors) or radiologist (deep tumors).
9. Prior chemotherapy or immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer: systemic or IT) must have been completed at least 4 weeks prior to dosing (with the exception of kinase inhibitors or other short half-life drugs, a 2 week washout is acceptable prior to treatment) and all adverse events have either returned to baseline or stabilized.

   Note: Subjects who have received prior platinum therapy are eligible irrespective of their response.
10. Prior systemic radiation therapy (either IV, intrahepatic or oral) completed at least 4 weeks prior to study drug administration; (for ipilimumab combination please see supplement FEC exclusion criteria).
11. Prior focal radiotherapy completed at least 2 weeks prior to study drug administration.
12. Prior major treatment-related surgery completed at least 4 weeks prior to study drug administration.
13. No prior primary or metastatic brain or meningeal tumors unless clinically and radiographically stable as well as off steroid therapy for at least 2 months.
14. Life expectancy ≥8 weeks; (for ipilimumab combination please see supplement FEC inclusion criteria).
15. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP)
    2. A WOCBP subject who may become pregnant or who are sexually active with a partner and who could become pregnant agrees to use an effective form of barrier contraception during the study and for at least 180 days in monotherapy; (for pembrolizumab and ipilimumab combinations please see supplements DEC/DEC2 and FEC for pregnancy criteria). (Male subjects must agree to use contraception and refrain from sperm donation during the study for 180 days after administration of study drug.)
16. Have adequate organ function as defined by the below screening laboratory values that must meet the following criteria:

    1. WBC ≥2000/μL (≥2 x 109/L).
    2. Neutrophils ≥1000/μL (≥1 x 109/L); (for pembrolizumab and ipilimumab combinations please see supplements DEC/DEC2 and FEC for neutrophil criteria).
    3. For subjects with planned superficial only injections: PT, PTT/aPTT, and INR ≤1.5 × ULN, Platelets ≥70x103/μL (≥ 70 x 109/L), Hemoglobin ≥8 g/dL
    4. Creatinine within the institution's laboratory upper limit of normal or calculated creatinine clearance >50 ml/min; (for pembrolizumab combination please see supplements DEC/DEC2 for creatine criteria).
    5. ALT (SGOT)/AST (SGPT) ≤2.5 x ULN without, and ≤ 5 x ULN with hepatic metastases.
    6. Bilirubin ≤2 x ULN (except subjects with Gilbert's syndrome, who must have total bilirubin <3.0 mg/dL (<52 µmol/L); (for pembrolizumab and ipilimumab combinations please see supplements DEC/DEC2 and FEC for bilirubin criteria).
    7. For subjects with planned deep tumor injections: PT, PTT/aPPT, and INR within normal limits; Platelet count ≥100,000/μL; hemoglobin ≥ 9 g/dL.

       Note: ALT (SGPT) =alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT) =aspartate aminotransferase (serum glutamic oxaloacetic transaminase); ULN=upper limit of normal.

       1 Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
17. Additional criteria for combination arms can be found in the appropriate combination protocol supplements. Refer to the Investigative site for details.

    Additional Inclusion Criteria for DEC2 cohort (anti-PD1 combination, KEYTRUDA® (pembrolizumab)) Population: Subjects with histologically or cytologically confirmed advanced or metastatic Pancreatic, Cholangiocarcinoma, non-MSI-H and/or MMR proficient colorectal cancer, and Squamous Cell Carcinoma tumors.

    Additional Inclusion Criteria for FEC cohort (anti-CTLA-4 combination, Yervoy (ipilimumab)) Population: Subjects with histologically or cytologically confirmed advanced or metastatic Hepatocellular carcinoma (HCC), breast cancer regardless of histology (BC) or soft tissue sarcoma

    NOTE: DEC and FEC combination cohorts have additional Inclusion Criteria - refer to the Investigative site for details.

    Exclusion Criteria:

    For INT230-6 Monotherapy cohort EC3, cohort DEC2-KEYTRUDA® combination and cohort FEC-Yervoy combination

    Subjects who exhibit any of the following conditions at screening will not be eligible for admission into the study:
18. History of severe hypersensitivity reactions to cisplatin or vinblastine or other products of the same class.
19. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or superficial bladder cancer, or any other cancer from which the subject has been disease-free for at least 2 years.
20. Subjects with tumors >15 cm (in longest diameter). Treatment plan for subjects with tumors that are 9 to15 cm must be discussed with and approved by the medical monitor.
21. Underlying medical condition that, in the Principal Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events.
22. Concurrent medical condition requiring the use of immunosuppressive medications, or systemic corticosteroids (topical steroids are permitted); systemic corticosteroids must be discontinued at least 4 weeks prior to dosing. Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if the subject is on a stable dose. Non-absorbed intra-articular steroid injections will be permitted; or use of other investigational drugs (drugs not marketed for any indication) within 30 days prior to study drug administration. Use of steroids as prophylactic treatment for subjects with contrast allergies to diagnostic imaging contrast dyes will be permitted.
23. For deep tumor cohorts, subjects who require uninterrupted anticoagulants of any type, on daily aspirin therapy or NSAIAs.
24. Use of other investigational drugs (drugs not marketed for any indication) within 28 days prior to study drug administration.

Pregnancy Exclusion:

A WOCBP who has a positive urine pregnancy test (e.g., within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

NOTE: DEC or FEC combination cohorts have additional Exclusion criteria. Refer to the Investigative site for details.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Schwartz, M.D., Study Director — Intensity Therapeutics; Lillian Siu, M.D., FRCP, Study Chair — Princess Margaret Hospital, Canada; Anthony El-Khoueiry, M.D., Principal Investigator — USC Norris and HOAG sites; Anthony J. Olszanski, M.D., RPh, Principal Investigator — Fox Chase Cancer Center; Nilofer Azad, M.D., Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Giles F Whalen, M.D., Principal Investigator — UMASS Memorial Medical Group; Matthew Ingham, M.D., Principal Investigator — Columbia University; Luis Camacho, M.D., Principal Investigator — Center for Oncology and Blood Disorders
Locations (8):
- United States (7):
  - USC Norris, Los Angeles, California
  - USC HOAG, Newport Beach, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Center for Oncology and Blood Disorders, Houston, Texas
- Princess Margaret Cancer Center - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One Subject (IT-004-016) had been enrolled in the study but deteriorated before the first dose was administered. The subject was originally planned to be placed in Cohort DEC2. This discontinuation means 110 patients were treated.
Groups:
- Monotherapy: Cohort A1: A1:INT230-6 injections every 28 days for 5 sessions into only superficial tumors, low starting dose, low concentration per tumor.
- Monotherapy: Cohort B1: B1:INT230-6 injections every 28 days for 5 sessions into deep tumors, low starting dose, low drug concentration per tumor Completed Cohort
- Monotherapy: Cohort EA: EA:INT230-6 injections every 2 weeks for 5 sessions into superficial tumors, medium starting dose, low drug concentration per tumor Completed Cohort
- Monotherapy: Cohort EC: EC:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, moderately high starting dose, high drug concentration per tumor Completed Cohort
- Monotherapy: Cohort EC-2: EC2:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, high starting dose, moderate drug concentration per tumor, higher number of tumors to be treated per session than EC.
- Monotherapy: Cohort EC3: EC3:INT230-6 injections every 2 weeks for 5 sessions at fixed maximal dose into superficial or deep tumors, unlimited number of tumors to be treated per session with retreatment once every 9 weeks for two years. Completed Cohort "
- INT 230-6 Combined With Pembrolizumab (Cohort DEC): DEC: INT230-6 injections every 2 weeks for 5 sessions with the possibility for INT230-6 retreatment into superficial tumors, with addition of anti-PD-1 antibody Keytruda (pembrolizumab) dosed concurrently starting at Day 1 every 3 weeks for two years for selected cancer types.
- INT 230-6 Combined With Pembrolizumab (Cohort DEC2): DEC2:INT230-6 per the dosing of cohort EC3 combined with Keytruda (pembrolizumab) dosed per DEC concurrently starting at Day 1 for selected cancers.
Period: Overall Study
Arm/Group | Monotherapy: Cohort A1 | Monotherapy: Cohort B1 | Monotherapy: Cohort EA | Monotherapy: Cohort EC | Monotherapy: Cohort EC-2 | Monotherapy: Cohort EC3 | INT 230-6 Combined With Pembrolizumab (Cohort DEC) | INT 230-6 Combined With Pembrolizumab (Cohort DEC2) | INT 230-6 Combined With Ipilimumab (Cohort FEC)
Started | 6 | 4 | 4 | 21 | 20 | 9 | 6 (2 Subjects (004-002 and 002-009) were originally treated on monotherapy (Cohorts EA and EC). They were later retreated on combination therapy with pembrolizumab in Cohort DEC. They will only be counted in participant flow once based on their original cohort assignment. The retreated subjects will be counted in their original and DEC for the adverse events section.) | 22 | 18
Completed | 1 | 1 | 1 | 9 | 9 | 3 | 3 | 5 | 13
Not Completed | 5 | 3 | 3 | 12 | 11 | 6 | 3 | 17 | 5
Not completed — Radiographic Deterioration | 0 | 3 | 1 | 2 | 6 | 3 | 0 | 4 | 2
Not completed — Adverse Event | 2 | 0 | 1 | 3 | 1 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 4 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 3 | 0
Not completed — Clinical Deterioration | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Refused Further Treatment | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Rapid Progression of Disease | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Monotherapy: (Cohort A1): A1:INT230-6 injections every 28 days for 5 sessions into only superficial tumors, low starting dose, low concentration per tumor.
- Monotherapy: (Cohort B1): B1:INT230-6 injections every 28 days for 5 sessions into deep tumors, low starting dose, low drug concentration per tumor Completed Cohort
- Monotherapy: (Cohort E-A): EA:INT230-6 injections every 2 weeks for 5 sessions into superficial tumors, medium starting dose, low drug concentration per tumor Completed Cohort
- Monotherapy: (Cohort E-C): EC:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, moderately high starting dose, high drug concentration per tumor Completed Cohort
- Monotherapy: (Cohort EC-2): EC2:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, high starting dose, moderate drug concentration per tumor, higher number of tumors to be treated per session than EC.
- Monotherapy: (Cohort EC3): EC3:INT230-6 injections every 2 weeks for 5 sessions at fixed maximal dose into superficial or deep tumors, unlimited number of tumors to be treated per session with retreatment once every 9 weeks for two years. Completed Cohort
- Total: Total of all reporting groups
Arm/Group | Monotherapy: (Cohort A1) | Monotherapy: (Cohort B1) | Monotherapy: (Cohort E-A) | Monotherapy: (Cohort E-C) | Monotherapy: (Cohort EC-2) | Monotherapy: (Cohort EC3) | INT 230-6 Combined With Pembrolizumab (Cohort DEC) | INT 230-6 Combined With Pembrolizumab (Cohort DEC2) | INT 230-6 Combined With Ipilimumab (Cohort FEC) | Total
Number analyzed (Participants) | 6 | 4 | 4 | 21 | 20 | 9 | 6 | 22 | 18 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 4 | 14 | 9 | 5 | 4 | 8 | 12 | 63
  >=65 years | 1 | 2 | 0 | 7 | 11 | 4 | 2 | 14 | 6 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (7.1) | 61.5 (7.9) | 57.6 (4.1) | 59.0 (9.9) | 64.6 (9.4) | 61.5 (11.3) | 64.2 (16) | 68.4 (7.3) | 64.2 (11.1) | 62.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 11 | 7 | 6 | 3 | 8 | 10 | 54
  Male | 2 | 1 | 2 | 10 | 13 | 3 | 3 | 14 | 8 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 3 | 3 | 13
  Not Hispanic or Latino | 6 | 4 | 3 | 19 | 18 | 7 | 6 | 19 | 15 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 3 | 2 | 2 | 1 | 5 | 1 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 7
  White | 5 | 3 | 4 | 16 | 18 | 5 | 5 | 13 | 13 | 82
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 0 | 0 | 1 | 1 | 0 | 4 | 1 | 1 | 11
  United States | 3 | 4 | 4 | 20 | 19 | 9 | 2 | 21 | 17 | 99

OUTCOME MEASURES:

1. Primary Outcome: Rate and Severity of Treatment-emergent Adverse Events ≥ Grade 3 Attributed to Study Drug Using the NCI Common Terminology Criteria for Adverse Events (CTCAE v.4.03) (Scale 1 to 5)
Description: The primary objective is to assess the safety and tolerability of single and multiple intratumoral doses of INT230-6 in subjects with advanced or recurrent malignancies. This will be assessed by the rate of ≥ grade 3 AE's attributed to INT230-6 and not the underlying disease.
  NCI Common Terminology Criteria for Adverse Events (CTCAE v.4.03) (Scale 1 (least severe) to 5 (most severe))
  All recorded adverse events will be listed and tabulated by system organ class, preferred term, and dose and coded according to the most current version of MedDRA. The incidence of adverse events will be tabulated and reviewed for potential significance and clinical importance.
  Adverse Events will be summarized for all reported data and by study period: a) up to and including 28 days post last dose of initial treatment, and b) from first dose of re-initiation of treatment, for subjects who re-initiate study therapy while in follow-up, up to 28 days post-dose of the last re-treatment dose.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy: Cohort A1 | Monotherapy: Cohort B1 | Monotherapy: Cohort EA | Monotherapy: Cohort EC | Monotherapy: Cohort EC-2 | Monotherapy: Cohort EC3 | INT 230-6 Combined With Pembrolizumab (Cohort DEC) | INT 230-6 Combined With Pembrolizumab (Cohort DEC2) | INT 230-6 Combined With Ipilimumab (Cohort FEC)
Number analyzed (Participants) | 6 | 4 | 4 | 21 | 20 | 9 | 6 | 22 | 18
Participants | 0 | 0 | 1 | 2 | 4 | 0 | 1 | 6 | 2

2. Secondary Outcome: Preliminary Efficacy: Assess the Preliminary Efficacy of INT230-6 by Measuring the Disease Control Rate (DCR) Based on the Response Evaluation Criteria in Solid Tumors (RECIST) and Immune RECIST (iRECIST) Criteria,
Description: Assess the preliminary efficacy of INT230-6 by measuring the disease control rate (CR+PR+SD) as assessed by iRECIST. Complete response (CR) and partial response (PR) will be defined for injected tumors followed per RECIST 1.1 utilizing target lesions. Progressive disease will be determined by clinical or radiological deterioration leading to the subject being taken off-treatment at the discretion of the investigator. Stable disease (SD) is defined as any adequate assessment not considered CR, PR, or progression.
Time Frame: Up to 5 years
Population: The cohorts A1/B1/EA/EC/EC2/EC3 were all "INT230-6 Monotherapy Treatment" and used to evaluate safety. DEC/DEC2 were "INT230-6+Pembrolizumab " were also used to evaluate safety. Per the Statistical Analysis Plan (SAP) the monotherapy cohorts were combined to evaluate efficacy in relation to total tumor burden (TTB) at doses of <40%TTB or ≥40%TTB for DCR. Per the SAP the pembrolizumab cohorts were combined to evaluate DCR.
Measure: Number; unit: percentage (DCR)
Groups:
- Monotherapy (Cohorts A1/B1/EA/EC/EC2/EC3) [Dosed >/= 40%TTB]: [This group was dosed >/= 40% of their Total Tumor Burden (TTB)]
  A1:INT230-6 injections every 28 days for 5 sessions into only superficial tumors, low starting dose, low concentration per tumor.
  Completed Cohort B1:INT230-6 injections every 28 days for 5 sessions into deep tumors, low starting dose, low drug concentration per tumor Completed Cohort EA:INT230-6 injections every 2 weeks for 5 sessions into superficial tumors, medium starting dose, low drug concentration per tumor Completed Cohort EC:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, moderately high starting dose, high drug concentration per tumor Completed Cohort EC2:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, high starting dose, moderate drug concentration per tumor, higher number of tumors to be treated per session than EC.
  Completed Cohort EC3:INT230-6 injections every 2 weeks for 5 sessions at fixed maximal dose into superficial or deep tumors, unlimited number of tumors to be treated per session with retreatment once every 9 weeks for two years. Completed Cohort
- Monotherapy (Cohorts A1/B1/EA/EC/EC2/EC3) [Dosed <40%TTB]: [This group was dosed <40% of their Total Tumor Burden (TTB)]
  A1:INT230-6 injections every 28 days for 5 sessions into only superficial tumors, low starting dose, low concentration per tumor.
  Completed Cohort B1:INT230-6 injections every 28 days for 5 sessions into deep tumors, low starting dose, low drug concentration per tumor Completed Cohort EA:INT230-6 injections every 2 weeks for 5 sessions into superficial tumors, medium starting dose, low drug concentration per tumor Completed Cohort EC:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, moderately high starting dose, high drug concentration per tumor Completed Cohort EC2:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, high starting dose, moderate drug concentration per tumor, higher number of tumors to be treated per session than EC.
  Completed Cohort EC3:INT230-6 injections every 2 weeks for 5 sessions at fixed maximal dose into superficial or deep tumors, unlimited number of tumors to be treated per session with retreatment once every 9 weeks for two years. Completed Cohort
Arm/Group | Monotherapy (Cohorts A1/B1/EA/EC/EC2/EC3) [Dosed >/= 40%TTB] | Monotherapy (Cohorts A1/B1/EA/EC/EC2/EC3) [Dosed <40%TTB] | INT230-6 Combined With Pembrolizumab (Cohorts DEC/DEC2) | INT 230-6 Combined With Ipilimumab (Cohort FEC)
Number analyzed (Participants) | 48 | 16 | 28 | 18
percentage (DCR) | 83.3 | 50.0 | 64.3 | 83.3

3. Secondary Outcome: Determine Pharmacokinetic Parameter Peak Plasma (Cmax in ng/mL) of Each of the 3 Main Components of INT230-6.
Description: Characterize the peak plasma profile for the three INT230-6 components after single and then multiple IT tumor site injections for safety purposes.
  Timepoints for sample collection were T = 1 Hours after dosing.
  Mean dose volume categories that were used to summarize data were as follows:
  2 mL (range 0 to 3.5 mL) 5 mL (range 3.6 to 6 mL) 10 mL (range >6 to 12 mL) 17 mL (range >12 to 24 mL) 30 mL (range >24 mL to 44 mL) 68 mL (range >44 to 98 mL) 118 mL (range >98 to 175 mL)
Time Frame: T = 1 hour after first dose
Population: The pharmacokinetic (PK) analysis aggregated subjects into groups by the dose given per convention according to our SAP and PK plan. Characterization of Patients who received similar doses (2mL, 5mL, 10mL, 18 mL, 30 mL, 68 mL, 118 mL, etc.) from all the cohorts were aggregated per the plan. This methodology of grouping (as described in the PK report produces meaningful API and excipient blood concentration profiles and determines conventional PK parameters for those agents.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pharmacokinetic (PK) Analysis Population (Component 1: Cisplatin): Pharmacokinetic analysis was conducted on 87 patients from the 110 treated. The population of 87 patients was based on available and detectable plasma concentration data. This group represents the PK data retrieved on the key component, Cisplatin.
- Pharmacokinetic Analysis Population (Component 2: SHAO): Pharmacokinetic Analysis was conducted on 87 patients from the 110 treated. The population of 87 patients was based on available and detectable plasma concentration data. This group represents the PK data retrieved on the key component, SHAO.
- Pharmacokinetic Analysis Population (Component 3: Vinblastine): Pharmacokinetic Analysis was conducted on 87 patients from the 110 treated. The population of 87 patients was based on available and detectable plasma concentration data. This group represents the PK data retrieved on the key component, Vinblastine.
Arm/Group | Pharmacokinetic (PK) Analysis Population (Component 1: Cisplatin) | Pharmacokinetic Analysis Population (Component 2: SHAO) | Pharmacokinetic Analysis Population (Component 3: Vinblastine)
Number analyzed (Participants) | 87 | 85 | 79
ng/mL
  Mean INT230-6 Dose Category: 2mL: number analyzed (Participants) | 10 | 8 | 3
  Mean INT230-6 Dose Category: 2mL | 34.27 (25.51) | 74.93 (70.8) | 1.35 (1.7)
  Mean INT230-6 Dose Category: 5mL: number analyzed (Participants) | 9 | 9 | 8
  Mean INT230-6 Dose Category: 5mL | 77.81 (38.16) | 113.7 (83.2) | .73 (.77)
  Mean INT230-6 Dose Category: 10mL: number analyzed (Participants) | 13 | 13 | 13
  Mean INT230-6 Dose Category: 10mL | 153.8 (65.75) | 300.6 (172.6) | .75 (.33)
  Mean INT230-6 Dose Category: 17mL: number analyzed (Participants) | 21 | 21 | 21
  Mean INT230-6 Dose Category: 17mL | 245.8 (119.3) | 426.8 (306.6) | 1.24 (.67)
  Mean INT230-6 Dose Category: 30mL: number analyzed (Participants) | 17 | 17 | 17
  Mean INT230-6 Dose Category: 30mL | 456.5 (195.0) | 911.6 (790.1) | 3.16 (1.99)
  Mean INT230-6 Dose Category: 68mL: number analyzed (Participants) | 13 | 13 | 13
  Mean INT230-6 Dose Category: 68mL | 952.2 (503.8) | 1446 (1245) | 5.63 (2.33)
  Mean INT230-6 Dose Category: 118mL: number analyzed (Participants) | 4 | 4 | 4
  Mean INT230-6 Dose Category: 118mL | 1673 (1276) | 2720 (1848) | 9.52 (4.52)

4. Secondary Outcome: Determine Key Pharmacokinetic Parameter, Area Under the Curve (AUC) (ng/mL) of Each of the 3 Main Components of INT230-6.
Description: Characterize the pharmacokinetic AUC profile of each of the three INT230-6 components for AUC after single IT tumor site injection for safety purposes.
  Timepoints for sample collection were T = 0, 1, 3, 6, 24 Hours after dosing.
  Mean dose volume categories that were used to summarize data were as follows:
  2 mL (range 0 to 3.5 mL) 5 mL (range 3.6 to 6 mL) 10 mL (range >6 to 12 mL) 17 mL (range >12 to 24 mL) 30 mL (range >24 mL to 44 mL) 68 mL (range >44 to 98 mL) 118 mL (range >98 to 175 mL)
Time Frame: T= 0, 1, 3, 6, 24 Hours after dosing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pharmacokinetic (PK) Analysis Population (Component 1: Cisplatin) | Pharmacokinetic Analysis Population (Component 2: SHAO) | Pharmacokinetic Analysis Population (Component 3: Vinblastine)
Number analyzed (Participants) | 87 | 85 | 79
ng/mL
  Mean INT230-6 Dose Category: 2mL Time point: 0 Hours: number analyzed (Participants) | 10 | 10 | 10
  Mean INT230-6 Dose Category: 2mL Time point: 0 Hours | 6.38 (20.18) | 0 (0) | .33 (1.05)
  Mean INT230-6 Dose Category: 2mL Time point: 1 Hour(s): number analyzed (Participants) | 10 | 10 | 10
  Mean INT230-6 Dose Category: 2mL Time point: 1 Hour(s) | 33.78 (24.92) | 59.94 (69.95) | .08 (.16)
  Mean INT230-6 Dose Category: 2mL Timepoint: 3 Hours: number analyzed (Participants) | 9 | 9 | 9
  Mean INT230-6 Dose Category: 2mL Timepoint: 3 Hours | 28.09 (23.16) | 3.33 (6.99) | .04 (.12)
  Mean INT230-6 Dose Category: 2mL Timepoint: 6 Hours: number analyzed (Participants) | 9 | 9 | 9
  Mean INT230-6 Dose Category: 2mL Timepoint: 6 Hours | 25.35 (20.35) | 0 (0) | 0 (0)
  Mean INT230-6 Dose Category: 2mL Timepoint: 24 Hours: number analyzed (Participants) | 10 | 10 | 10
  Mean INT230-6 Dose Category: 2mL Timepoint: 24 Hours | 20.74 (17.22) | 0 (0) | 0 (0)
  Mean INT230-6 Dose Category: 5mL Timepoint: 0 Hours: number analyzed (Participants) | 9 | 9 | 9
  Mean INT230-6 Dose Category: 5mL Timepoint: 0 Hours | 1.56 (4.67) | 0 (0) | 0 (0)
  Mean INT230-6 Dose Category: 5mL Timepoint: 1 Hour(s): number analyzed (Participants) | 9 | 9 | 9
  Mean INT230-6 Dose Category: 5mL Timepoint: 1 Hour(s) | 77.81 (38.16) | 113.74 (83.23) | .65 (.76)
  Mean INT230-6 Dose Category: 5mL Timepoint: 3 Hours: number analyzed (Participants) | 9 | 8 | 9
  Mean INT230-6 Dose Category: 5mL Timepoint: 3 Hours | 58.50 (30.57) | 11.43 (15.52) | .16 (.16)
  Mean INT230-6 Dose Category: 5mL Timepoint: 6 Hours: number analyzed (Participants) | 9 | 8 | 9
  Mean INT230-6 Dose Category: 5mL Timepoint: 6 Hours | 59.04 (32.03) | 2.18 (6.15) | 0 (0)
  Mean INT230-6 Dose Category: 5mL Timepoint: 24 Hours: number analyzed (Participants) | 9 | 8 | 8
  Mean INT230-6 Dose Category: 5mL Timepoint: 24 Hours | 53.87 (29.07) | 0 (0) | 0 (0)
  Mean INT230-6 Dose Category: 10mL Timepoint: 0 Hours: number analyzed (Participants) | 13 | 13 | 13
  Mean INT230-6 Dose Category: 10mL Timepoint: 0 Hours | 4.95 (13.09) | 0 (0) | 0 (0)
  Mean INT230-6 Dose Category: 10mL Timepoint: 1 Hour(s): number analyzed (Participants) | 13 | 13 | 13
  Mean INT230-6 Dose Category: 10mL Timepoint: 1 Hour(s) | 152.63 (67.36) | 300.56 (172.62) | .74 (.35)
  Mean INT230-6 Dose Category: 10mL Timepoint: 3 Hours: number analyzed (Participants) | 13 | 13 | 13
  Mean INT230-6 Dose Category: 10mL Timepoint: 3 Hours | 114.7 (53.38) | 36.68 (51.13) | .39 (.22)
  Mean INT230-6 Dose Category: 10mL Timepoint: 6 Hours: number analyzed (Participants) | 12 | 12 | 12
  Mean INT230-6 Dose Category: 10mL Timepoint: 6 Hours | 111.57 (49.37) | 6.21 (15.22) | .34 (.1)
  Mean INT230-6 Dose Category: 10mL Timepoint: 24 Hours: number analyzed (Participants) | 13 | 13 | 12
  Mean INT230-6 Dose Category: 10mL Timepoint: 24 Hours | 100.98 (52.36) | 0 (0) | .05 (.12)
  Mean INT230-6 Dose Category: 17mL Timepoint: 0 Hours: number analyzed (Participants) | 21 | 21 | 21
  Mean INT230-6 Dose Category: 17mL Timepoint: 0 Hours | 4.99 (19.50) | 0 (0) | .01 (.06)
  Mean INT230-6 Dose Category: 17mL Timepoint: 1 Hours: number analyzed (Participants) | 21 | 21 | 21
  Mean INT230-6 Dose Category: 17mL Timepoint: 1 Hours | 233.15 (125.77) | 426.75 (306.59) | 1.2 (.72)
  Mean INT230-6 Dose Category: 17mL Timepoint: 3 Hours: number analyzed (Participants) | 21 | 21 | 21
  Mean INT230-6 Dose Category: 17mL Timepoint: 3 Hours | 187.08 (93.22) | 59.76 (45.33) | .66 (.35)
  Mean INT230-6 Dose Category: 17mL Timepoint: 6 Hours: number analyzed (Participants) | 21 | 85 | 21
  Mean INT230-6 Dose Category: 17mL Timepoint: 6 Hours | 176.45 (90.26) | 19.49 (19.77) | .51 (.29)
  Mean INT230-6 Dose Category: 17mL Timepoint:24 Hours: number analyzed (Participants) | 21 | 21 | 21
  Mean INT230-6 Dose Category: 17mL Timepoint:24 Hours | 163.87 (90.19) | .5 (2.27) | .17 (.24)
  Mean INT230-6 Dose Category: 30mL Timepoint: 0 Hours: number analyzed (Participants) | 17 | 17 | 17
  Mean INT230-6 Dose Category: 30mL Timepoint: 0 Hours | 7.15 (19.24) | 0.0 (0) | 0 (0)
  Mean INT230-6 Dose Category: 30mL Timepoint: 1 Hours: number analyzed (Participants) | 17 | 17 | 17
  Mean INT230-6 Dose Category: 30mL Timepoint: 1 Hours | 456.47 (195.02) | 911.55 (790.14) | 3.16 (1.99)
  Mean INT230-6 Dose Category: 30mL Timepoint: 3 Hours: number analyzed (Participants) | 17 | 17 | 17
  Mean INT230-6 Dose Category: 30mL Timepoint: 3 Hours | 344.82 (163.12) | 95.67 (64.38) | 1.44 (.77)
  Mean INT230-6 Dose Category: 30mL Timepoint: 6 Hours: number analyzed (Participants) | 16 | 16 | 16
  Mean INT230-6 Dose Category: 30mL Timepoint: 6 Hours | 325.73 (152.91) | 26.95 (20.34) | 1.06 (.58)
  Mean INT230-6 Dose Category: 30mL Timepoint: 24 Hours: number analyzed (Participants) | 17 | 17 | 17
  Mean INT230-6 Dose Category: 30mL Timepoint: 24 Hours | 295.42 (137.46) | .78 (3.20) | .47 (.38)
  Mean INT230-6 Dose Category: 68mL Timepoint: 0 Hours: number analyzed (Participants) | 13 | 13 | 13
  Mean INT230-6 Dose Category: 68mL Timepoint: 0 Hours | 62.93 (222.70) | 289.23 (1042.84) | .44 (1.58)
  Mean INT230-6 Dose Category: 68mL Timepoint: 1 Hours: number analyzed (Participants) | 13 | 13 | 13
  Mean INT230-6 Dose Category: 68mL Timepoint: 1 Hours | 832.92 (192.93) | 1286.00 (1039.43) | 5.53 (2.35)
  Mean INT230-6 Dose Category: 68mL Timepoint: 3 Hours: number analyzed (Participants) | 13 | 13 | 13
  Mean INT230-6 Dose Category: 68mL Timepoint: 3 Hours | 741.92 (343.37) | 240.82 (276.13) | 2.73 (.72)
  Mean INT230-6 Dose Category: 68mL Timepoint: 6 Hours: number analyzed (Participants) | 12 | 12 | 12
  Mean INT230-6 Dose Category: 68mL Timepoint: 6 Hours | 775.00 (581.44) | 96.54 (146.88) | 1.94 (.55)
  Mean INT230-6 Dose Category: 68mL Timepoint: 24 Hours: number analyzed (Participants) | 13 | 12 | 13
  Mean INT230-6 Dose Category: 68mL Timepoint: 24 Hours | 610.08 (264.39) | 2.71 (6.44) | .94 (.43)
  Mean INT230-6 Dose Category: 118mL Timepoint: 0 Hours: number analyzed (Participants) | 4 | 4 | 4
  Mean INT230-6 Dose Category: 118mL Timepoint: 0 Hours | 0 (0) | 0 (0) | .08 (.17)
  Mean INT230-6 Dose Category: 118mL Timepoint: 1 Hours: number analyzed (Participants) | 4 | 4 | 4
  Mean INT230-6 Dose Category: 118mL Timepoint: 1 Hours | 1664 (1287.53) | 2719.75 (1848.17) | 9.52 (4.52)
  Mean INT230-6 Dose Category: 118mL Timepoint: 3 Hours: number analyzed (Participants) | 3 | 3 | 3
  Mean INT230-6 Dose Category: 118mL Timepoint: 3 Hours | 875 (433.39) | 459.67 (289.46) | 4.33 (1.46)
  Mean INT230-6 Dose Category: 118mL Timepoint: 6 Hours: number analyzed (Participants) | 3 | 3 | 3
  Mean INT230-6 Dose Category: 118mL Timepoint: 6 Hours | 779.67 (360.88) | 183.43 (99.64) | 3.08 (.85)
  Mean INT230-6 Dose Category: 118mL Timepoint: 24 Hours: number analyzed (Participants) | 3 | 3 | 3
  Mean INT230-6 Dose Category: 118mL Timepoint: 24 Hours | 945.33 (544.78) | 21.93 (24.84) | 1.24 (1.19)

5. Secondary Outcome: Key Pharmacokinetic Parameters, Half Live (Hours) of Each of the 3 Main Components of INT230-6.
Description: Characterize the half life of each of the three INT230-6 components after single and multiple IT tumor site injections for safety purposes.
  Timepoints for sample collection were T = 0, 1, 3, 6, 24 Hours after dosing.
  Mean dose volume categories that were used to summarize data were as follows:
  2 mL (range 0 to 3.5 mL) 5 mL (range 3.6 to 6 mL) 10 mL (range >6 to 12 mL) 17 mL (range >12 to 24 mL) 30 mL (range >24 mL to 44 mL) 68 mL (range >44 to 98 mL) 118 mL (range >98 to 175 mL)
Time Frame: T= 0, 1, 3, 6, 24 hours
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pharmacokinetic (PK) Analysis Population (Component 1: Cisplatin) | Pharmacokinetic Analysis Population (Component 2: SHAO) | Pharmacokinetic Analysis Population (Component 3: Vinblastine)
Number analyzed (Participants) | 26 | 6 | 28
Hours
  Mean INT230-6 Dose Category: 2mL: number analyzed (Participants) | 4 | 0 | 0
  Mean INT230-6 Dose Category: 2mL | 77.98 (34.92) |  |
  Mean INT230-6 Dose Category: 5mL: number analyzed (Participants) | 4 | 0 | 0
  Mean INT230-6 Dose Category: 5mL | 130.4 (129.8) |  |
  Mean INT230-6 Dose Category: 10mL: number analyzed (Participants) | 3 | 0 | 1
  Mean INT230-6 Dose Category: 10mL | 106.3 (53.58) |  | 18.82
  Mean INT230-6 Dose Category: 17mL: number analyzed (Participants) | 5 | 1 | 6
  Mean INT230-6 Dose Category: 17mL | 78.73 (66.36) | 7.33 | 20.11 (7.45)
  Mean INT230-6 Dose Category: 30mL: number analyzed (Participants) | 7 | 1 | 10
  Mean INT230-6 Dose Category: 30mL | 64.77 (15.18) | 7.48 | 15.35 (4.38)
  Mean INT230-6 Dose Category: 68mL: number analyzed (Participants) | 3 | 3 | 9
  Mean INT230-6 Dose Category: 68mL | 129.4 (125.5) | 3.91 (2.6) | 14.06 (3.7)
  Mean INT230-6 Dose Category: 118mL: number analyzed (Participants) | 0 | 1 | 28
  Mean INT230-6 Dose Category: 118mL |  | 6.18 | 24.48 (4.76)

6. Other Pre Specified Outcome: Exploratory: Control or Regression of Non Injected Tumors by Measurement of Length (in Centimeters) Radio-graphically Using Computer Tomography or Magnetic Resonance Imaging.
Description: Characterize response in non-injected lesions (up to 5) using length (cm) as the key parameter for measurement.
Time Frame: Up to 18 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Exploratory: Blood, Genetic and Tissue Biomarker Identification From Cell Flow Phenotyping, Tissue Analysis, Genetic SNP Analysis.
Description: Evaluate various tumor and anti-tumor immune response biomarkers from blood, tumor tissue that may correlate with tumor response. Flow and tissue panels may include Live-Dead, CD3, CD4, CD8, FoxP3, Ki-67, ICOS, DAPI, PD-1, LAG-3, TIM-3, CTLA-4 and analysis of blood serum cytokine such as Th1/Th2, IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12 p70, IL-13, and TNF-α.
Time Frame: Up to 2 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Exploratory: Overall Subject Outcome
Description: Evaluate overall response by iRECIST including survival
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Each patient would have their Adverse Events recorded starting at the first dose until 28 days after the last dose. up to 5 years.
Groups:
- Monotherapy: (Cohort A1): A1:INT230-6 injections every 28 days for 5 sessions into only superficial tumors, low starting dose, low concentration per tumor.
  Completed Cohort
- Monotherapy: (Cohort EC-2): EC2:INT230-6 injections every 2 weeks for 5 sessions into superficial or deep tumors, high starting dose, moderate drug concentration per tumor, higher number of tumors to be treated per session than EC.
  Completed Cohort
- INT230-6 Combined With Pembrolizumab (Cohorts DEC): DEC: INT230-6 injections every 2 weeks for 5 sessions with the possibility for INT230-6 retreatment into superficial tumors, with addition of anti-PD-1 antibody KEYTRUDA® (pembrolizumab) dosed concurrently starting at Day 1 every 3 weeks for two years for selected cancer types.
  Completed Cohort
- INT230-6 Combined With Pembrolizumab (Cohorts DEC2): DEC2:INT230-6 per the dosing of cohort EC3 combined with KEYTRUDA® (pembrolizumab) dosed per DEC concurrently starting at Day 1 for selected cancers.
Arm/Group | Monotherapy: (Cohort A1) | Monotherapy: (Cohort B1) | Monotherapy: (Cohort E-A) | Monotherapy: (Cohort E-C) | Monotherapy: (Cohort EC-2) | Monotherapy: (Cohort EC3) | INT230-6 Combined With Pembrolizumab (Cohorts DEC) | INT230-6 Combined With Pembrolizumab (Cohorts DEC2) | INT 230-6 Combined With Ipilimumab (Cohort FEC)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/4 | 0/21 | 0/20 | 0/9 | 0/8 | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/4 | 1/21 | 1/20 | 1/9 | 2/8 | 2/22 | 1/18
Other Adverse Events (participants affected / at risk) | 4/6 | 2/4 | 3/4 | 20/21 | 20/20 | 7/9 | 7/8 | 19/22 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: (Cohort A1) (N=6) | Monotherapy: (Cohort B1) (N=4) | Monotherapy: (Cohort E-A) (N=4) | Monotherapy: (Cohort E-C) (N=21) | Monotherapy: (Cohort EC-2) (N=20) | Monotherapy: (Cohort EC3) (N=9) | INT230-6 Combined With Pembrolizumab (Cohorts DEC) (N=8) | INT230-6 Combined With Pembrolizumab (Cohorts DEC2) (N=22) | INT 230-6 Combined With Ipilimumab (Cohort FEC) (N=18)
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localized Tumor Related Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: (Cohort A1) (N=6) | Monotherapy: (Cohort B1) (N=4) | Monotherapy: (Cohort E-A) (N=4) | Monotherapy: (Cohort E-C) (N=21) | Monotherapy: (Cohort EC-2) (N=20) | Monotherapy: (Cohort EC3) (N=9) | INT230-6 Combined With Pembrolizumab (Cohorts DEC) (N=8) | INT230-6 Combined With Pembrolizumab (Cohorts DEC2) (N=22) | INT 230-6 Combined With Ipilimumab (Cohort FEC) (N=18)
Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localized Tumor-Related Pain (General disorders) | 2 | 2 | 3 | 13 | 14 | 6 | 5 | 10 | 9
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 11 | 10 | 5 | 2 | 2 | 4
Fatigue (General disorders) | 1 | 0 | 0 | 11 | 8 | 0 | 0 | 6 | 6
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7 | 7 | 1 | 1 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 10 | 6 | 1 | 3 | 3 | 3
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Injection Site Erythema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 6 | 0 | 0 | 2 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
Injection Site Induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection Site Odema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Distention (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 4 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 3
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Parathesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Tumor Necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pruritus Genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gamma-Glutamyl Transferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Axillary Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection Site Bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Upper Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmer Plantar Erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling Face (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swollen Tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT03058289/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT03058289/SAP_001.pdf